CLINICAL TRIAL: NCT05481957
Title: Clinical Efficacy and Safety of Vortioxetine Combined With Mood Stabilizer in the Treatment of Bipolar Disorder Type II Depression
Brief Title: Vortioxetine Adjunctive Treatment in Bipolar Depression
Acronym: Vortioxetine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu ShaoHua, Department of Psychiatry, First Affiliated Hospital of Zhejiang University, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20210111C-R1
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Vortioxetine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vortioxetine (Experimental): participants given 5~10mg per day for 16 weeks
  Interventions: Drug: Vortioxetine
- Sodium valproate (Active Comparator): participants given 500~1000mg per day for 16 weeks
  Interventions: Drug: valprote

INTERVENTIONS:
Drug: Vortioxetine — 5-10mg for 16 weeks
  Other Names: Brintellix®
  Arms: vortioxetine
Drug: valprote — 500~1000mg for 16 weeks
  Other Names: Depakine
  Arms: Sodium valproate

SUMMARY:
Depressive episode of bipolar disorder is often the first symptom of patients with bipolar disorder, which is characterized by frequent recurrence, relatively long duration, high comorbidity rate and high fatality rate. People with bipolar disorder spend a third of their lives depressed, and it is these depressive symptoms that lead to long-term disability and early death. The treatment of bipolar depression is controversial. The latest Mood Disorders CPG guidelines recommend first-line therapy: quetiapine, lurasidone, lithium, valproate, lamotrigine monotherapy or combination of quetiapine, lurasidone plus Mood stabilizer, olanzapine plus fluoxetine therapy. In addition, the use of antidepressants is still controversial, and their efficacy, prognosis and risk of mania remain to be evaluated. Vortioxetine is a novel antidepressant with unique characteristics, and its multi-mode mechanism of action can be used to treat a wide spectrum of symptoms of depression. Current clinical experience suggests that the clinical conversion rate of vortioxetine is low, and the depressive symptoms and cognitive symptoms of people with depressive episodes are significantly improved. As of September 2019, a total of 4.87 million patient years (nearly 3 months of treatment with 20 million patients) were treated with vortioxetine in PSUR (Periodic Safety Update), with 51 reported cases of hypomania and 322 reported cases of mania. Based on the above data, the post-marketing conversion rate of vortioxetine is approximately 1 in 10,000 patient-years or 1 in 40,000 patients. Therefore, the efficacy and risk of transferring to mania of vortioxetine in bipolar II depressive episode deserve further investigation.

DETAILED DESCRIPTION:
This study initiated by The first affiliated hospital of zhejiang university. Professor Shao-hua Hu will be PI of the study. There are about 80 patients with bipolar II depressive episode were involved in this study, all participants after 4 weeks of monotherapy (quetiapine or lurasidone). Group A: Those patients who were treated effectively over the 4th weekend {Reduction rate of 17 items of the Hamilton Depression Scale (HDS-17) >50%} continued with the original regimen for 4 weeks. Subjects who did not meet valid criteria (HSDRS-17 subscore ratio<50%) were randomly assigned to two treatment groups: group B (quetiapine/lurasidone + vortioxetine tablets) and group C (quetiapine/lurasidone + sodium valproate sustained release tablets). Subjects in group B were given vortioxetine in combination with their original treatment regimen at week 5; Subjects in group C began to receive sodium valproate sustained-release tablets in combination with the original treatment regimen at week 5. All three groups were observed at the end of the 16th week.

Group A: single drug treatment group: quetiapine tablet 300mg~600mg/d or Lurasidone tablet 40-120mg /d; Group B: quetiapine tablets 300mg~600mg/d or Lurasidone tablets 40-120mg /d+ vortioxetine 5-10mg /d Group C: quetiapine tablets 300mg~600mg/d or Lurasidone tablets 40-120mg /d+ sodium valproate sustained release tablets 0.5-1.0 /d Quetiapine or lurasidone is currently the first-line treatment for bipolar II depressive episodes, ensuring effective treatment for all subjects. The study program will last 16 weeks with seven study visits including screening. For the consideration of scientific, legal and ethical factors, 100 subjects are initially planned to be enrolled in this experiment.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between >18.5 and <29.5 kg
2. The MINI-International Neuropsychiatric Interview is adopted and patients selected shall meet the clinical diagnostic criteria stipulated in DSM-5 on clinical diagnostic criteria for type II bipolar depression.
3. HDRS17>17
4. YMRS score <5;
5. No treatment was given before enrollment;
6. All patients and their family members were informed and agreed to this trial.

Exclusion Criteria:

1. Those who suffering from other severe mental diseases;
2. Those who suffering from severe somatic diseases;
3. Those who had received medication (such as anti-depressants, antipsychotics, mood stabilizers, etc.) within 1 month before enrollment;
4. Those who had been treated with ECT one month before enrollment;
5. Those who currently have severe suicidal thoughts or behavior, or who are extremely excited and fail to cooperate with;
6. Women in pregnancy and lactation;
7. Patients with contraindications to drugs used in this trial;
8. Those who have participated in a clinical trial of an investigational product in the last 60 days

10) Substance misuse/abuse

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 131 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale(MADRS) | 0 ~16 weeks
  Montgomery-Asberg Depression Rating Scale(MADRS) score is to evaluate the degree of depression, and the higher score means severer depression. Score frame: 0~60. The higher score means severer depression.

CONTACTS AND LOCATIONS:
Overall Officials: Li YouMing, Study Chair — Zhejiang University
Locations (1):
- Department of Psychiatry, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Arms and interventions can be shared, while the clinical data will not be shared